CLINICAL TRIAL: NCT03678233
Title: Efficacy of Testosterone Gel to Restore Normal Serum Values of Testosterone During the Acute Phase of Critical Illness in Adult ICU Patients
Acronym: TestICUs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-404; 2017-004978-34 (Other: 2017-004978-34)
Record Dates: First submitted 2018-09-03; First posted 2018-09-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hypermetabolism in ICU; Loss of Muscle Mass; Functional Disability After ICU; ICU Acquired Hypogonadism; Treatment With Testosterone Gel in ICU
Keywords: hypermetabolism; hypogonadism; testosterone
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): AndroGel® AndroGel 16.2 mg/L will be applied to upper arms or shoulders once a day at 9:00 am to dry and intact skin for a period of 28 days or until ICU discharge. The daily dose 101.25 mg in men and 20.25 mg in women
  Interventions: Drug: AndroGel 16.2 mg/L
- Control (No Intervention): In the control group, AndroGel will not be administered.

INTERVENTIONS:
Drug: AndroGel 16.2 mg/L — Testosterone gel 1.62 % will be applied to upper arms or shoulders once a day at 9:00 am to dry and intact skin for a period of 28 days or until ICU discharge. The daily dose 101.25 mg in men and 20.25 mg in women.
  Arms: Intervention

SUMMARY:
Critically ill patients experience major insults that lead to increased protein catabolism. Hypermetabolism occurs early and rapidly during the first week of critical illness to provide amino acids for the production of energy via gluconeogenesis, and also for the synthesis of acute phase proteins and repair of tissue damage. During acute phase, neuroendocrine and inflammatory responses promote protein breakdown and amino acid release. Under stress conditions, protein synthesis cannot match the increased rate of muscle proteolysis because of a state of anabolism resistance, which limits uptake of amino acids into muscles. Hypermetabolism results in a significant loss of lean body mass with an impact on weaning from the ventilator and muscle recovery. Functional disability may be long term sometimes with no full return to normal.

In critically ill patients, severe and persistent testosterone deficiency is very common and is observed early after ICU admission. This acquired hypogonadism promotes the persistent loss of skeletal muscle protein and is related to poor outcome.

Administration of testosterone induces skeletal muscle fiber hypertrophy, decreases protein breakdown in healthy young men and burned patients. It has been repeatedly shown that testosterone treatment enhances muscle mass and strength in young and older hypogonadal men and women and can improve physical performance.

DETAILED DESCRIPTION:
Type of trial

TestICUs-1 is a single center open-label parallel randomized controlled study phase II assessing the efficacy of testosterone gel to correct low testosterone serum levels associated with ICU acquired hypogonadism in mechanically ventilated patients with shock. TestICUs-1 will be conducted in the 10-bed medical ICU of the university hospital of Clermont-Ferrand. Study drug is Androgel® 1.62 mg/L approved by the ANSM for the treatment of hypogonadism in men containing 1.62% of testosterone.

Category of research Research involving human subjects aimed at assessing the efficacy of and safety to drug.

Study phase

* II/ Feasibility
* Technology Readiness Level : 7 B

A study assessing the efficacy of a multimodal strategy including treatment with testosterone gel, (75 mg/day in men and 25 mg/day in women) in improving physical activity in hemodialysis patients is in progress (Americano PHRC N 2012, AE Heng).

ELIGIBILITY:
Inclusion Criteria:

* - Males and females aged over 18 years receiving invasive mechanical ventilation
* Invasive mechanical ventilation expected to be required for more than 48 hours
* Treatment with vasoactive drugs
* Written informed consent obtained from the legal representative
* Social security cover

Exclusion Criteria:

* - History of prostate or breast cancer, prostatic specific antigen (PSA) ≥ 4 ng/ml
* ICU length of stay > 72 h before enrollment
* Moribund defined as having a score SAPS II > 75 12 hours after admission
* Pre-existing illness with a life expectancy of <6 months
* Cardiac arrest
* Preexistent cognitive impairment or language barrier
* Acute intracranial or spinal cord injury
* Acute hemorrhagic or ischemic stroke
* Neuromuscular disease (Guillain-Barré, myasthenia)
* Inability to walk without assistance prior to acute ICU illness (use of a cane or walkers not excluded)
* Documented allergy to testosterone
* Age > 80 years
* Pregnancy or breast feeding
* Patient on judicial protection

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pourcentage of patients with normal median value of serum total testosterone | day 4 to day 14
  Pourcentage of patients with median value of serum total testosterone collected from blood samples at day 4, 7, 10, 14 higher than 280 ng/dl in men and 12 ng/dl in women.

SECONDARY OUTCOMES:
Proportion of patients with normal median free testosterone serum values | day 4 to day 14
  Proportion of patients with median free testosterone serum values at day 4, 7, 10, 14 higher than 58 pg/ml in men and 0,9 ng/ml in women
Proportion of patients with normal median serum values of bioavailable testosterone | day 4 to day 14
  Proportion of patients with median serum values of bioavailable testosterone at day 4, 7, 10, 14 higher than 75 ng/dl in men 0.8 ng/dl in women
Nitrogen balance | daily from day 1 to day 14
  Daily and cumulative nitrogen balance from day 1 to extubation
Physical performance | day 14, 1month and 3 months after ICU discharge
  Physical performance by Six-minute walk test (6MWT)
Muscle strength | at ICU discharge, 1month and 3 months after ICU discharge
  Muscle strength by MRC (Medical Research Scale)
Near Infrared Spectroscopy | at 14 days
  Near Infrared Spectroscopy by NIRS test
Muscular mass | at ICU discharge and 1month after ICU discharge
  Muscular mass by L3 computed tomography
Lung function | at 1 and 3 months after ICU discharge
  Lung function by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos BACHOUMAS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Plank LD, Connolly AB, Hill GL. Sequential changes in the metabolic response in severely septic patients during the first 23 days after the onset of peritonitis. Ann Surg. 1998 Aug;228(2):146-58. doi: 10.1097/00000658-199808000-00002. PMID 9712558
- [Background] Hussain SN, Mofarrahi M, Sigala I, Kim HC, Vassilakopoulos T, Maltais F, Bellenis I, Chaturvedi R, Gottfried SB, Metrakos P, Danialou G, Matecki S, Jaber S, Petrof BJ, Goldberg P. Mechanical ventilation-induced diaphragm disuse in humans triggers autophagy. Am J Respir Crit Care Med. 2010 Dec 1;182(11):1377-86. doi: 10.1164/rccm.201002-0234OC. Epub 2010 Jul 16. PMID 20639440
- [Background] Vanhorebeek I, Gunst J, Derde S, Derese I, Boussemaere M, Guiza F, Martinet W, Timmermans JP, D'Hoore A, Wouters PJ, Van den Berghe G. Insufficient activation of autophagy allows cellular damage to accumulate in critically ill patients. J Clin Endocrinol Metab. 2011 Apr;96(4):E633-45. doi: 10.1210/jc.2010-2563. Epub 2011 Jan 26. PMID 21270330
- [Background] Weijs PJ, Cynober L, DeLegge M, Kreymann G, Wernerman J, Wolfe RR. Proteins and amino acids are fundamental to optimal nutrition support in critically ill patients. Crit Care. 2014 Nov 17;18(6):591. doi: 10.1186/s13054-014-0591-0. PMID 25565377
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Dos Santos C, Hussain SN, Mathur S, Picard M, Herridge M, Correa J, Bain A, Guo Y, Advani A, Advani SL, Tomlinson G, Katzberg H, Streutker CJ, Cameron JI, Schols A, Gosker HR, Batt J; MEND ICU Group; RECOVER Program Investigators; Canadian Critical Care Translational Biology Group. Mechanisms of Chronic Muscle Wasting and Dysfunction after an Intensive Care Unit Stay. A Pilot Study. Am J Respir Crit Care Med. 2016 Oct 1;194(7):821-830. doi: 10.1164/rccm.201512-2344OC. PMID 27058306
- [Background] Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, Ali NA, Sharshar T. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37(10 Suppl):S299-308. doi: 10.1097/CCM.0b013e3181b6ef67. PMID 20046114
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Fletcher SN, Kennedy DD, Ghosh IR, Misra VP, Kiff K, Coakley JH, Hinds CJ. Persistent neuromuscular and neurophysiologic abnormalities in long-term survivors of prolonged critical illness. Crit Care Med. 2003 Apr;31(4):1012-6. doi: 10.1097/01.CCM.0000053651.38421.D9. PMID 12682465
- [Background] Solverson KJ, Grant C, Doig CJ. Assessment and predictors of physical functioning post-hospital discharge in survivors of critical illness. Ann Intensive Care. 2016 Dec;6(1):92. doi: 10.1186/s13613-016-0187-8. Epub 2016 Sep 20. PMID 27646108
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Ma L, Shen C, Chai J, Yin H, Deng H, Feng R. Extracellular signal-regulated kinase-mammalian target of rapamycin signaling and forkhead-box transcription factor 3a phosphorylation are involved in testosterone's effect on severe burn injury in a rat model. Shock. 2015 Jan;43(1):85-91. doi: 10.1097/SHK.0000000000000244. PMID 25057926
- [Background] Ferrando AA, Sheffield-Moore M, Yeckel CW, Gilkison C, Jiang J, Achacosa A, Lieberman SA, Tipton K, Wolfe RR, Urban RJ. Testosterone administration to older men improves muscle function: molecular and physiological mechanisms. Am J Physiol Endocrinol Metab. 2002 Mar;282(3):E601-7. doi: 10.1152/ajpendo.00362.2001. PMID 11832363
- [Background] Snyder PJ, Peachey H, Hannoush P, Berlin JA, Loh L, Lenrow DA, Holmes JH, Dlewati A, Santanna J, Rosen CJ, Strom BL. Effect of testosterone treatment on body composition and muscle strength in men over 65 years of age. J Clin Endocrinol Metab. 1999 Aug;84(8):2647-53. doi: 10.1210/jcem.84.8.5885. PMID 10443654
- [Background] Diaz EC, Herndon DN, Porter C, Sidossis LS, Suman OE, Borsheim E. Effects of pharmacological interventions on muscle protein synthesis and breakdown in recovery from burns. Burns. 2015 Jun;41(4):649-57. doi: 10.1016/j.burns.2014.10.010. Epub 2014 Nov 16. PMID 25468473
- [Background] Bhasin S, Woodhouse L, Casaburi R, Singh AB, Bhasin D, Berman N, Chen X, Yarasheski KE, Magliano L, Dzekov C, Dzekov J, Bross R, Phillips J, Sinha-Hikim I, Shen R, Storer TW. Testosterone dose-response relationships in healthy young men. Am J Physiol Endocrinol Metab. 2001 Dec;281(6):E1172-81. doi: 10.1152/ajpendo.2001.281.6.E1172. PMID 11701431
- [Background] Sinha-Hikim I, Artaza J, Woodhouse L, Gonzalez-Cadavid N, Singh AB, Lee MI, Storer TW, Casaburi R, Shen R, Bhasin S. Testosterone-induced increase in muscle size in healthy young men is associated with muscle fiber hypertrophy. Am J Physiol Endocrinol Metab. 2002 Jul;283(1):E154-64. doi: 10.1152/ajpendo.00502.2001. PMID 12067856
- [Background] Sinha-Hikim I, Roth SM, Lee MI, Bhasin S. Testosterone-induced muscle hypertrophy is associated with an increase in satellite cell number in healthy, young men. Am J Physiol Endocrinol Metab. 2003 Jul;285(1):E197-205. doi: 10.1152/ajpendo.00370.2002. Epub 2003 Apr 1. PMID 12670837
- [Background] Brodsky IG, Balagopal P, Nair KS. Effects of testosterone replacement on muscle mass and muscle protein synthesis in hypogonadal men--a clinical research center study. J Clin Endocrinol Metab. 1996 Oct;81(10):3469-75. doi: 10.1210/jcem.81.10.8855787.
- [Background] Urban RJ, Bodenburg YH, Gilkison C, Foxworth J, Coggan AR, Wolfe RR, Ferrando A. Testosterone administration to elderly men increases skeletal muscle strength and protein synthesis. Am J Physiol. 1995 Nov;269(5 Pt 1):E820-6. doi: 10.1152/ajpendo.1995.269.5.E820. PMID 7491931
- [Background] Ferrando AA, Sheffield-Moore M, Wolf SE, Herndon DN, Wolfe RR. Testosterone administration in severe burns ameliorates muscle catabolism. Crit Care Med. 2001 Oct;29(10):1936-42. doi: 10.1097/00003246-200110000-00015. PMID 11588456
- [Background] Liva SM, Voskuhl RR. Testosterone acts directly on CD4+ T lymphocytes to increase IL-10 production. J Immunol. 2001 Aug 15;167(4):2060-7. doi: 10.4049/jimmunol.167.4.2060. PMID 11489988
- [Background] Khosla S, Atkinson EJ, Dunstan CR, O'Fallon WM. Effect of estrogen versus testosterone on circulating osteoprotegerin and other cytokine levels in normal elderly men. J Clin Endocrinol Metab. 2002 Apr;87(4):1550-4. doi: 10.1210/jcem.87.4.8397. PMID 11932280
- [Background] Malkin CJ, Pugh PJ, Jones RD, Kapoor D, Channer KS, Jones TH. The effect of testosterone replacement on endogenous inflammatory cytokines and lipid profiles in hypogonadal men. J Clin Endocrinol Metab. 2004 Jul;89(7):3313-8. doi: 10.1210/jc.2003-031069. PMID 15240608
- [Background] Tsilidis KK, Rohrmann S, McGlynn KA, Nyante SJ, Lopez DS, Bradwin G, Feinleib M, Joshu CE, Kanarek N, Nelson WG, Selvin E, Platz EA. Association between endogenous sex steroid hormones and inflammatory biomarkers in US men. Andrology. 2013 Nov;1(6):919-28. doi: 10.1111/j.2047-2927.2013.00129.x. Epub 2013 Sep 30. PMID 24124163
- [Background] Zhang Y, Gao Y, Tan A, Yang X, Zhang H, Zhang S, Wu C, Lu Z, Wang M, Liao M, Qin X, Li L, Hu Y, Mo Z. Endogenous sex hormones and C-reactive protein in healthy Chinese men. Clin Endocrinol (Oxf). 2013 Jan;78(1):60-6. doi: 10.1111/j.1365-2265.2012.04359.x. PMID 22313436
- [Background] Sharshar T, Bastuji-Garin S, De Jonghe B, Stevens RD, Polito A, Maxime V, Rodriguez P, Cerf C, Outin H, Touraine P, Laborde K. Hormonal status and ICU-acquired paresis in critically ill patients. Intensive Care Med. 2010 Aug;36(8):1318-26. doi: 10.1007/s00134-010-1840-6. Epub 2010 Mar 24. PMID 20333354
- [Background] Vogel AV, Peake GT, Rada RT. Pituitary-testicular axis dysfunction in burned men. J Clin Endocrinol Metab. 1985 Apr;60(4):658-65. doi: 10.1210/jcem-60-4-658. PMID 4038713
- [Background] Wang C, Chan V, Yeung RT. Effect of surgical stress on pituitary-testicular function. Clin Endocrinol (Oxf). 1978 Sep;9(3):255-66. doi: 10.1111/j.1365-2265.1978.tb02208.x. PMID 361300
- [Background] Van den Berghe G, de Zegher F, Lauwers P, Veldhuis JD. Luteinizing hormone secretion and hypoandrogenaemia in critically ill men: effect of dopamine. Clin Endocrinol (Oxf). 1994 Nov;41(5):563-9. doi: 10.1111/j.1365-2265.1994.tb01819.x. PMID 7828343
- [Background] Nierman DM, Mechanick JI. Hypotestosteronemia in chronically critically ill men. Crit Care Med. 1999 Nov;27(11):2418-21. doi: 10.1097/00003246-199911000-00016. PMID 10579258
- [Background] Kim JJ, Oh SJ, Shin JH, Hwang SY, Hyun SY, Yang HJ, Lee G. Testosterone related good neurologic outcome on the patients with return of spontaneous circulation after cardiac arrest: a prospective cohort study. Resuscitation. 2013 May;84(5):645-50. doi: 10.1016/j.resuscitation.2012.10.022. Epub 2012 Nov 7. PMID 23142200
- [Background] Bhasin S, Storer TW, Berman N, Yarasheski KE, Clevenger B, Phillips J, Lee WP, Bunnell TJ, Casaburi R. Testosterone replacement increases fat-free mass and muscle size in hypogonadal men. J Clin Endocrinol Metab. 1997 Feb;82(2):407-13. doi: 10.1210/jcem.82.2.3733. PMID 9024227
- [Background] Wang C, Swerdloff RS, Iranmanesh A, Dobs A, Snyder PJ, Cunningham G, Matsumoto AM, Weber T, Berman N; Testosterone Gel Study Group. Transdermal testosterone gel improves sexual function, mood, muscle strength, and body composition parameters in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2839-53. doi: 10.1210/jcem.85.8.6747. PMID 10946892
- [Background] Bhasin S, Woodhouse L, Casaburi R, Singh AB, Mac RP, Lee M, Yarasheski KE, Sinha-Hikim I, Dzekov C, Dzekov J, Magliano L, Storer TW. Older men are as responsive as young men to the anabolic effects of graded doses of testosterone on the skeletal muscle. J Clin Endocrinol Metab. 2005 Feb;90(2):678-88. doi: 10.1210/jc.2004-1184. Epub 2004 Nov 23. PMID 15562020
- [Background] Storer TW, Basaria S, Traustadottir T, Harman SM, Pencina K, Li Z, Travison TG, Miciek R, Tsitouras P, Hally K, Huang G, Bhasin S. Effects of Testosterone Supplementation for 3 Years on Muscle Performance and Physical Function in Older Men. J Clin Endocrinol Metab. 2017 Feb 1;102(2):583-593. doi: 10.1210/jc.2016-2771. PMID 27754805
- [Background] Snyder PJ, Peachey H, Berlin JA, Hannoush P, Haddad G, Dlewati A, Santanna J, Loh L, Lenrow DA, Holmes JH, Kapoor SC, Atkinson LE, Strom BL. Effects of testosterone replacement in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2670-7. doi: 10.1210/jcem.85.8.6731. PMID 10946864
- [Background] Sheffield-Moore M, Paddon-Jones D, Casperson SL, Gilkison C, Volpi E, Wolf SE, Jiang J, Rosenblatt JI, Urban RJ. Androgen therapy induces muscle protein anabolism in older women. J Clin Endocrinol Metab. 2006 Oct;91(10):3844-9. doi: 10.1210/jc.2006-0588. Epub 2006 Aug 8. PMID 16895962
- [Background] Miller KK, Biller BM, Beauregard C, Lipman JG, Jones J, Schoenfeld D, Sherman JC, Swearingen B, Loeffler J, Klibanski A. Effects of testosterone replacement in androgen-deficient women with hypopituitarism: a randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2006 May;91(5):1683-90. doi: 10.1210/jc.2005-2596. Epub 2006 Feb 14. PMID 16478814
- [Background] Miller BE, De Souza MJ, Slade K, Luciano AA. Sublingual administration of micronized estradiol and progesterone, with and without micronized testosterone: effect on biochemical markers of bone metabolism and bone mineral density. Menopause. 2000 Sep-Oct;7(5):318-26. doi: 10.1097/00042192-200007050-00006. PMID 10993031
- [Background] Davis SR, McCloud P, Strauss BJ, Burger H. Testosterone enhances estradiol's effects on postmenopausal bone density and sexuality. Maturitas. 1995 Apr;21(3):227-36. doi: 10.1016/0378-5122(94)00898-h. PMID 7616872
- [Background] Chapman IM, Visvanathan R, Hammond AJ, Morley JE, Field JB, Tai K, Belobrajdic DP, Chen RY, Horowitz M. Effect of testosterone and a nutritional supplement, alone and in combination, on hospital admissions in undernourished older men and women. Am J Clin Nutr. 2009 Mar;89(3):880-9. doi: 10.3945/ajcn.2008.26538. Epub 2009 Jan 14. PMID 19144729
- [Background] White HD, Brown LA, Gyurik RJ, Manganiello PD, Robinson TD, Hallock LS, Lewis LD, Yeo KT. Treatment of pain in fibromyalgia patients with testosterone gel: Pharmacokinetics and clinical response. Int Immunopharmacol. 2015 Aug;27(2):249-56. doi: 10.1016/j.intimp.2015.05.016. Epub 2015 May 21. PMID 26004317
- [Background] Bhasin S, Storer TW, Javanbakht M, Berman N, Yarasheski KE, Phillips J, Dike M, Sinha-Hikim I, Shen R, Hays RD, Beall G. Testosterone replacement and resistance exercise in HIV-infected men with weight loss and low testosterone levels. JAMA. 2000 Feb 9;283(6):763-70. doi: 10.1001/jama.283.6.763. PMID 10683055
- [Background] Bhasin S, Storer TW, Asbel-Sethi N, Kilbourne A, Hays R, Sinha-Hikim I, Shen R, Arver S, Beall G. Effects of testosterone replacement with a nongenital, transdermal system, Androderm, in human immunodeficiency virus-infected men with low testosterone levels. J Clin Endocrinol Metab. 1998 Sep;83(9):3155-62. doi: 10.1210/jcem.83.9.5079. PMID 9745419
- [Background] Johansen KL, Mulligan K, Schambelan M. Anabolic effects of nandrolone decanoate in patients receiving dialysis: a randomized controlled trial. JAMA. 1999 Apr 14;281(14):1275-81. doi: 10.1001/jama.281.14.1275. PMID 10208142
- [Background] Schols AM, Soeters PB, Mostert R, Pluymers RJ, Wouters EF. Physiologic effects of nutritional support and anabolic steroids in patients with chronic obstructive pulmonary disease. A placebo-controlled randomized trial. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1268-74. doi: 10.1164/ajrccm.152.4.7551381.
- [Background] Casaburi R, Bhasin S, Cosentino L, Porszasz J, Somfay A, Lewis MI, Fournier M, Storer TW. Effects of testosterone and resistance training in men with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Oct 15;170(8):870-8. doi: 10.1164/rccm.200305-617OC. Epub 2004 Jul 21. PMID 15271690
- [Background] Li H, Guo Y, Yang Z, Roy M, Guo Q. The efficacy and safety of oxandrolone treatment for patients with severe burns: A systematic review and meta-analysis. Burns. 2016 Jun;42(4):717-27. doi: 10.1016/j.burns.2015.08.023. Epub 2015 Oct 9. PMID 26454425
- [Background] Gervasio JM, Dickerson RN, Swearingen J, Yates ME, Yuen C, Fabian TC, Croce MA, Brown RO. Oxandrolone in trauma patients. Pharmacotherapy. 2000 Nov;20(11):1328-34. doi: 10.1592/phco.20.17.1328.34889. PMID 11079282
- [Background] Bulger EM, Jurkovich GJ, Farver CL, Klotz P, Maier RV. Oxandrolone does not improve outcome of ventilator dependent surgical patients. Ann Surg. 2004 Sep;240(3):472-8; discussion 478-80. doi: 10.1097/01.sla.0000137131.22608.e2. PMID 15319718
- [Background] Shoskes JJ, Wilson MK, Spinner ML. Pharmacology of testosterone replacement therapy preparations. Transl Androl Urol. 2016 Dec;5(6):834-843. doi: 10.21037/tau.2016.07.10. PMID 28078214
- [Background] Yoshida EM, Erb SR, Scudamore CH, Owen DA. Severe cholestasis and jaundice secondary to an esterified testosterone, a non-C17 alkylated anabolic steroid. J Clin Gastroenterol. 1994 Apr;18(3):268-70. doi: 10.1097/00004836-199404000-00036. No abstract available. PMID 8034945
- [Background] Jeschke MG, Finnerty CC, Suman OE, Kulp G, Mlcak RP, Herndon DN. The effect of oxandrolone on the endocrinologic, inflammatory, and hypermetabolic responses during the acute phase postburn. Ann Surg. 2007 Sep;246(3):351-60; discussion 360-2. doi: 10.1097/SLA.0b013e318146980e. PMID 17717439
- [Background] Dobs AS, Meikle AW, Arver S, Sanders SW, Caramelli KE, Mazer NA. Pharmacokinetics, efficacy, and safety of a permeation-enhanced testosterone transdermal system in comparison with bi-weekly injections of testosterone enanthate for the treatment of hypogonadal men. J Clin Endocrinol Metab. 1999 Oct;84(10):3469-78. doi: 10.1210/jcem.84.10.6078. PMID 10522982
- [Background] Ullah MI, Riche DM, Koch CA. Transdermal testosterone replacement therapy in men. Drug Des Devel Ther. 2014 Jan 9;8:101-12. doi: 10.2147/DDDT.S43475. eCollection 2014. PMID 24470750
- [Background] Dillon EL, Durham WJ, Urban RJ, Sheffield-Moore M. Hormone treatment and muscle anabolism during aging: androgens. Clin Nutr. 2010 Dec;29(6):697-700. doi: 10.1016/j.clnu.2010.03.010. Epub 2010 May 7. PMID 20452103
- [Background] Basaria S, Coviello AD, Travison TG, Storer TW, Farwell WR, Jette AM, Eder R, Tennstedt S, Ulloor J, Zhang A, Choong K, Lakshman KM, Mazer NA, Miciek R, Krasnoff J, Elmi A, Knapp PE, Brooks B, Appleman E, Aggarwal S, Bhasin G, Hede-Brierley L, Bhatia A, Collins L, LeBrasseur N, Fiore LD, Bhasin S. Adverse events associated with testosterone administration. N Engl J Med. 2010 Jul 8;363(2):109-22. doi: 10.1056/NEJMoa1000485. Epub 2010 Jun 30. PMID 20592293
- [Background] Vigen R, O'Donnell CI, Baron AE, Grunwald GK, Maddox TM, Bradley SM, Barqawi A, Woning G, Wierman ME, Plomondon ME, Rumsfeld JS, Ho PM. Association of testosterone therapy with mortality, myocardial infarction, and stroke in men with low testosterone levels. JAMA. 2013 Nov 6;310(17):1829-36. doi: 10.1001/jama.2013.280386. PMID 24193080
- [Background] Finkle WD, Greenland S, Ridgeway GK, Adams JL, Frasco MA, Cook MB, Fraumeni JF Jr, Hoover RN. Increased risk of non-fatal myocardial infarction following testosterone therapy prescription in men. PLoS One. 2014 Jan 29;9(1):e85805. doi: 10.1371/journal.pone.0085805. eCollection 2014. PMID 24489673
- [Background] Snyder PJ, Bhasin S, Cunningham GR, Matsumoto AM, Stephens-Shields AJ, Cauley JA, Gill TM, Barrett-Connor E, Swerdloff RS, Wang C, Ensrud KE, Lewis CE, Farrar JT, Cella D, Rosen RC, Pahor M, Crandall JP, Molitch ME, Cifelli D, Dougar D, Fluharty L, Resnick SM, Storer TW, Anton S, Basaria S, Diem SJ, Hou X, Mohler ER 3rd, Parsons JK, Wenger NK, Zeldow B, Landis JR, Ellenberg SS; Testosterone Trials Investigators. Effects of Testosterone Treatment in Older Men. N Engl J Med. 2016 Feb 18;374(7):611-24. doi: 10.1056/NEJMoa1506119. PMID 26886521
- [Background] Basaria S, Harman SM, Travison TG, Hodis H, Tsitouras P, Budoff M, Pencina KM, Vita J, Dzekov C, Mazer NA, Coviello AD, Knapp PE, Hally K, Pinjic E, Yan M, Storer TW, Bhasin S. Effects of Testosterone Administration for 3 Years on Subclinical Atherosclerosis Progression in Older Men With Low or Low-Normal Testosterone Levels: A Randomized Clinical Trial. JAMA. 2015 Aug 11;314(6):570-81. doi: 10.1001/jama.2015.8881. PMID 26262795
- [Background] English KM, Steeds RP, Jones TH, Diver MJ, Channer KS. Low-dose transdermal testosterone therapy improves angina threshold in men with chronic stable angina: A randomized, double-blind, placebo-controlled study. Circulation. 2000 Oct 17;102(16):1906-11. doi: 10.1161/01.cir.102.16.1906. PMID 11034937
- [Background] Baillargeon J, Urban RJ, Kuo YF, Ottenbacher KJ, Raji MA, Du F, Lin YL, Goodwin JS. Risk of Myocardial Infarction in Older Men Receiving Testosterone Therapy. Ann Pharmacother. 2014 Sep;48(9):1138-1144. doi: 10.1177/1060028014539918. Epub 2014 Jul 2. PMID 24989174
- [Background] Corona G, Maseroli E, Rastrelli G, Isidori AM, Sforza A, Mannucci E, Maggi M. Cardiovascular risk associated with testosterone-boosting medications: a systematic review and meta-analysis. Expert Opin Drug Saf. 2014 Oct;13(10):1327-51. doi: 10.1517/14740338.2014.950653. Epub 2014 Aug 19. PMID 25139126
- [Background] Borst SE, Shuster JJ, Zou B, Ye F, Jia H, Wokhlu A, Yarrow JF. Cardiovascular risks and elevation of serum DHT vary by route of testosterone administration: a systematic review and meta-analysis. BMC Med. 2014 Nov 27;12:211. doi: 10.1186/s12916-014-0211-5. PMID 25428524
- [Background] Davis SR, Moreau M, Kroll R, Bouchard C, Panay N, Gass M, Braunstein GD, Hirschberg AL, Rodenberg C, Pack S, Koch H, Moufarege A, Studd J; APHRODITE Study Team. Testosterone for low libido in postmenopausal women not taking estrogen. N Engl J Med. 2008 Nov 6;359(19):2005-17. doi: 10.1056/NEJMoa0707302. PMID 18987368
- [Background] Singh AB, Lee ML, Sinha-Hikim I, Kushnir M, Meikle W, Rockwood A, Afework S, Bhasin S. Pharmacokinetics of a testosterone gel in healthy postmenopausal women. J Clin Endocrinol Metab. 2006 Jan;91(1):136-44. doi: 10.1210/jc.2005-1640. Epub 2005 Nov 1. PMID 16263817
- [Background] Mackenzie TA, Clark NG, Bistrian BR, Flatt JP, Hallowell EM, Blackburn GL. A simple method for estimating nitrogen balance in hospitalized patients: a review and supporting data for a previously proposed technique. J Am Coll Nutr. 1985;4(5):575-81. doi: 10.1080/07315724.1985.10720100. PMID 3932497
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Muscular weakness assessment: use of normal isometric strength data. The National Isometric Muscle Strength (NIMS) Database Consortium. Arch Phys Med Rehabil. 1996 Dec;77(12):1251-5. doi: 10.1016/s0003-9993(96)90188-4. PMID 8976307
- [Background] Dyer C. US authorities face legal challenges over anaesthetics used in executions. BMJ. 2011 Mar 24;342:d1925. doi: 10.1136/bmj.d1925. No abstract available. PMID 21436110
- [Background] Ryan TE, Brophy P, Lin CT, Hickner RC, Neufer PD. Assessment of in vivo skeletal muscle mitochondrial respiratory capacity in humans by near-infrared spectroscopy: a comparison with in situ measurements. J Physiol. 2014 Aug 1;592(15):3231-41. doi: 10.1113/jphysiol.2014.274456. Epub 2014 Jun 20. PMID 24951618
- [Background] Adami A, Cao R, Porszasz J, Casaburi R, Rossiter HB. Reproducibility of NIRS assessment of muscle oxidative capacity in smokers with and without COPD. Respir Physiol Neurobiol. 2017 Jan;235:18-26. doi: 10.1016/j.resp.2016.09.008. Epub 2016 Sep 19. PMID 27659351
- [Background] Mourtzakis M, Prado CM, Lieffers JR, Reiman T, McCargar LJ, Baracos VE. A practical and precise approach to quantification of body composition in cancer patients using computed tomography images acquired during routine care. Appl Physiol Nutr Metab. 2008 Oct;33(5):997-1006. doi: 10.1139/H08-075. PMID 18923576
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863